CLINICAL TRIAL: NCT03200769
Title: Study of the Efficacy of the Treatment of Sleep Apnea Syndrome by CPAP in Pharmacoresistant Epilepsy
Acronym: SASER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012_66; 2013-A01156-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-06-12; First posted 2017-06-27 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Sleep Apnea Syndromes; Epilepsies, Partial
Keywords: CPAP; Sleep Apnea Syndrome; Pharmacoresistant Epilepsy; Apnea Hypopnea-Index
MeSH Terms: conditions — Sleep Apnea Syndromes; Epilepsies, Partial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group I (No Intervention): AHI/h < 15
- Group IIa (Experimental): 15 < AHI/h < 30. Randomization group. Intervention : CPAP active
  Interventions: Device: CPAP active
- Group IIb (Experimental): 15 < AHI/h < 30. Randomization group. Intervention : CPAP placebo during the first 3 months. After this period, the patient will have the possibility to continue with an active CPAP.
  Interventions: Device: CPAP placebo
- Group III (Active Comparator): AHI/h > 30. Intervention : CPAP active
  Interventions: Device: CPAP active

INTERVENTIONS:
Device: CPAP active — CPAP PR1 Philips Respironics with a pression between 4 and 14 mm Hg
  Arms: Group III; Group IIa
Device: CPAP placebo — CPAP PR1 Philips Respironics with a constant pression of 4 mm Hg.
  Arms: Group IIb

SUMMARY:
Study of the Efficacy of the Treatment of Sleep Apnea Syndrome by CPAP in Pharmacoresistant Epilepsy. The primary goal is to evaluate the efficacity after 3 months of obstructive sleep apnea syndrome treatment by CPAP on the epilepsy seizures frequency.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18.
* Patient suffering of pharmacoresistant epilepsy.
* Frequency of epilepsy crisis : minimum 4 per month.
* Antiepileptic drug on a stable dose for at least 2 months.
* SA-SDQ score ≥ 25.
* Written informed consent obtained.
* Patient affiliated with a social security regimen.

Exclusion Criteria:

* Pregnant females (female subjects who are lactating are not excluded).
* Anterior CPAP treatment.
* Central apnea >20% during the initial polysomnography.
* Mental retardation or severe cognitive impairment.
* Presence of pseudo-crisis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Number of patients from group IIa and IIb with decreased seizure frequency | At 3 months
  Decreased > 50% after CPAP treatment

SECONDARY OUTCOMES:
Number of patients from group IIa and IIb with decreased seizure frequency | At 6 months ; At 12 months
  Decreased > 50% after CPAP treatment
Number of patients from group III with decreased seizure frequency | At 3 months ; At 6 months ; At 12 months
  Decreased > 50% after CPAP treatment
Impact of AHI on the number of night seizures | At 12 months
  Does the AHI has an impact on the number of night seizure?
Impact of the localisation and the type of epilepsy based on patient medical history exam (video-electroencephalogram) on the SAS risk | At 12 months
  Does the AHI is impacted by the localisation and the type of epilepsy?
Number of seizures based on the seizures diary | At 12 months
  Impact of SAS treatment on the pharmacoresistance
Number of patients who became drug-susceptible based on the seizures diary | At 3 months ; At 6 months ; At 12 months
  Impact of SAS treatment on the pharmacoresistance
Quality of life questionnaire (QOLIE 31) | At 3 months ; At 6 months ; At 12 months
  Impact of SAS treatment on the quality of life
Anxiety and depression questionnaire (BECK) | At 3 months ; At 6 months ; At 12 months
  Impact of SAS treatment on anxiety and depression
Somnolence questionnaire (Epworth) | At 3 months ; At 6 months ; At 12 months
  Impact of SAS treatment on somnolence
Cognitive capacity questionnaire (MOCA) | At 3 months ; At 6 months ; At 12 months
  Impact of SAS treatment on cognitive capacity questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DERAMBURE, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU de Lille - Rue Emile LAINE - Hopitâl Roger Salengro Rez de Chaussée - Neurophysiologie Clinique, Lille, France